CLINICAL TRIAL: NCT01322737
Title: Evaluation of a Novel Endoscopic Polypectomy Device in Excised Human Colon and Gastric Tissue.
Brief Title: Feasibility Trial to Evaluate the Ability of the SuMO Tissue Access and Resection System
Acronym: SUMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Apollo Endosurgery, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, Director, Surgical Endoscopy, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 06-10-21
Record Dates: First submitted 2011-03-07; First posted 2011-03-25 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Colon Disease; Gastric Disease
Keywords: resection; open; laparoscopic; benign; malignant; disease; colon; gastric
MeSH Terms: conditions — Colonic Diseases; Stomach Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SUMO Tissue Access and Resection System (Experimental)
  Interventions: Procedure: Tissue Access and Resection System

INTERVENTIONS:
Procedure: Tissue Access and Resection System — This feasibility trial will assess the effectiveness of SuMO System to create a submucosal pocket and resect the overlying mucosa in excised human colonic or gastric tissue
  Other Names: SUMO Tissue Access and Resection System

SUMMARY:
This feasibility trial will evaluate the ability of the SuMO Tissue Access and Resection System (Apollo Endosurgery, Austin, Texas). The SuMO System utilizes balloons to create a submucosal pocket and electrosurgical cutting device to resect the mucosa. The SuMO elevates the tissue from the underlying muscularis using a balloon to distend the submucosa, similar to what is currently performed with injectable saline in a standard EMR. After dissection of the lesion, a separate cutting device will be utilized to resect the tissue by cutting around the border of the targeted tissue. If needed, a standard loop snare will be used to complete the mucosal resection.

DETAILED DESCRIPTION:
The subject will already be scheduled for segmental colectomy or gastrectomy.

The colectomy or gastrectomy specimen will be prepared on a side table for an ex vivo endoscopic procedure. The ends of the stomach or colon, if not already stapled closed will be ligated to allow for insufflation. The endoscope will be placed into the excised organ and the SuMO System devices will be deployed away from any areas of excised pathologic tissue, so as not to disrupt the pathologist's evaluation of the excised tissue. The specimen will then be opened and grossly examined for the actual completeness of the submucosal pocket and resection. Mucosal and muscular wall disruptions will be assessed. Again, no interference in the underlying pathology will be performed. If sufficient specimen is present, the SuMO procedure may be repeated on the same specimen.

Following the performance of the EMR by the SUMO balloon system on the ex vivo colon specimen, both the resected piece of tissue and the site of resection will be evaluated pathologically by H and E staining. Specifically, the depth of resection in the ex vivo colon specimen will be determined. In addition, the level of dissection on the removed piece of mucosa will also be identified.

During this procedure still images or a video recording maybe captured, however all images will be taken of the removed specimen. There will not be any patient identifiers on any of the images or DVD's taken during the procedure.

No clinical follow up is required, as the treated area will have already been resected and there is no risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Established indication for open or laparoscopic or colon resection or gastrectomy
* Subject agrees to participate, fully understands content of informed consent form, and signs the informed consent form

Exclusion Criteria:

* Subjects that are minors or prisoners
* Subjects who would have difficulty comprehending or complying with the requirements of the study
* Subjects who fail to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evidence of the ability of the SUMO device to create a submucosal pocket and resect the overlying mucosa in human colon or stomach. | (day one)The colon or stomach tissue is evaluated in the Operating Room immediatley following excision. Subjects are not followed after using the excised tissue in the operating room.
  Assess the feasibility of the SuMO device for creation of a submucosal pocket and resecting the overlying mucosa in a segment of excised human colon or stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Marks, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States